CLINICAL TRIAL: NCT04063904
Title: Pilot Study of an Ambulatory Medical Abortion Service at 13-18 Weeks of Gestation in Colombia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties with recruitment, COVID 19 pandemic
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1044
Record Dates: First submitted 2019-08-13; First posted 2019-08-21 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Second Trimester Abortion
Keywords: medical abortion; mifepristone
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mifepristone and misoprostol (Experimental): Mifepristone 200 mg orally, followed 24-48 hours later by misoprostol 400mcg sublingually every three hours until the abortion occurs. The experimental part of the regimen is that the first dose of misoprostol will be taken 1-2 hours before arriving at the clinic for continued dosing, monitoring and abortion completion.
  Interventions: Drug: Mifepristone; Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — One 200 mg pill (oral)
Drug: Misoprostol — Two 400 mcg pills (sublingual)

SUMMARY:
This pilot study seeks to evaluate the safety, acceptability and feasibility of a shortened outpatient procedure for medical abortion at 13-18 weeks gestation. It also seeks to document the roles of health workers in providing services related to later abortion care. Participants will take a single dose of 200 mg mifepristone orally, followed 24-48 hours later with 400 mcg misoprostol sublingually prior to arriving at the study clinic. Repeat doses of 400 mcg misoprostol will be administered sublingually every three hours at the clinic until the abortion is achieved. If expulsion does not occur by a certain time prior to the clinic closing that day, D&E will be performed to complete the abortion.

ELIGIBILITY:
Inclusion Criteria:

1. Have an intrauterine pregnancy of 13-18 weeks gestation according to ultrasound
2. Meet legal criteria to obtain abortion
3. Be at least 18 years old
4. Have access to a phone where she can be reached for the 2-week follow up
5. Be willing to follow pilot study procedures

Exclusion Criteria:

1. Known allergy to mifepristone or misoprostol/prostaglandin or other contraindications to the use of mifepristone or misoprostol
2. Any contraindications to vaginal delivery
3. More than one prior cesarean delivery
4. Staying more than 2 hours away from the clinic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2021-04-03 (Actual)

PRIMARY OUTCOMES:
Successful medical abortion | 0-60 hours after mifepristone
  Proportion of women who have a successful abortion with medication only and are discharged from care on the same day as misoprostol induction.

SECONDARY OUTCOMES:
Induction-to-abortion interval | 0-12 hours after misoprostol
  Time (median min/hrs) from first misoprostol dose until fetal and placental expulsion
Initiation-to-abortion interval | 0-60 hours after mifepristone
  Time (median min/hrs) from mifepristone administration until fetal and placental expulsion
Total dose of misoprostol administered | 0-12 hours after misoprostol
  Mean number of misoprostol doses administered to achieve abortion
Method safety | Two weeks after mifepristone
  Proportion of participants who experience: extramural delivery, hemorrhage requiring transfusion, infection, uterine rupture, prolonged hospitalization, any complications
Tasks performed by clinic staff | From enrollment through discharge from care (approx. 3 days)
  Type of task performed (i.e. counseling, monitoring vital signs, administering drugs, monitoring woman's condition, post-abortion contraception, managing discharge) per cadre of provider
Total clinic time | 0-12 hours from arrival at clinic on day of induction with misoprostol
  Time (median hrs) since arrival to clinic on day of misoprostol dosing to discharge from care that same day
Pain with procedure | 0-12 hours after first misoprostol dose
  Mean pain score (scale 0-10)
Side effects | 0-12 hours after first misoprostol dose
  Report of side effects and proportion of participants who experienced each one
Satisfaction with procedure | Prior to discharge from care on day of abortion, up to 12 hours after first misoprostol dose
  Proportion of participants who reported the procedure as satisfactory or very satisfactory

CONTACTS AND LOCATIONS:
Overall Officials: Ilana G Dzuba, MHS, Principal Investigator — Gynuity Health Projects; Maria Mercedes Vivas, MD, Principal Investigator — Fundacion Orientame; Juliette Ortiz, Study Director — Fundacion Orientame; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (1):
- Fundacion Orientame, Bogotá, Colombia